CLINICAL TRIAL: NCT02782143
Title: Testing the Validity of the "Modified Confusion Assessment Method for the Emergency Department" (mCAM-ED)" for the Recognition of Delirium in Elderly Patient Admitted to the Emergency Department
Brief Title: Testing the Validity of the "Modified Confusion Assessment Method for the Emergency Department" (mCAM-ED)"
Acronym: Val_mCAM-ED
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ-2015-123
Record Dates: First submitted 2015-12-16; First posted 2016-05-25 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Delirium
Keywords: delirium detection
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed Study validates the accuracy of the modified Confusion Assessment Method for the Emergency Department

DETAILED DESCRIPTION:
Delirium is a complex neuropsychiatric syndrome with sudden change in cognition such as disturbance in orientation or memory particularly in elderly patients in the context of acute illness. Multiple complications such as falls or increased duration of hospitalisation may result in delirium. Long-term consequences may result in increased mortality rates and higher admissions rates to nursing homes. In 2012, delirium prevalence in the Emergency Department (ED) of the University Hospital Basel was 9.5% in patients with 65 years and over. Although a systematic delirium management was introduced in 2012, without systematic screening delirium detection rates varies between 20 and 40% only. The risk of non-detection over the complete hospitalisation is high when early delirium detection did not occur in the ED. In a preliminary evaluation we could show the usefulness of the mCAM-ED

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years

Exclusion Criteria:

* patients under resuscitation or fatal illness
* not speaking German
* being aphasic
* being deaf

Ages: 65 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients admitted to the emergency department being 65 years and over
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Delirium measured by geriatricians using Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria | once during the stay at the emergency department which lasts an average of 24 hours
  acute confusional states in patients
Delirium measured by geriatricians using DSM-5 criteria | once during the stay at the emergency department which lasts an average of 24 hours
  acute confusional states in patients
Delirium measured by advanced practice nurses using the mCAM-ED | once during the stay at the emergency department which lasts an average of 24 hours
  acute confusional states in patients
degree of concordance between nurses' delirium measurement versus geriatricians' delirium measurement assessed in a four field matrix | once during the stay at the emergency department which lasts an average of 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hasemann, PhD, Study Chair — usb
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Background] Trzepacz, P. T., & Meagher, D. J. (2008). Neuropsychiatric Aspects of Delirium. In S. C. Yudofsky & R. E. Hales (Eds.), Neuropsychiatry and Behavioral Neurosciences (5 ed., pp. 445-518). Washington, DC: American Psychiatric Publishing, Inc.
- [Background] Han JH, Zimmerman EE, Cutler N, Schnelle J, Morandi A, Dittus RS, Storrow AB, Ely EW. Delirium in older emergency department patients: recognition, risk factors, and psychomotor subtypes. Acad Emerg Med. 2009 Mar;16(3):193-200. doi: 10.1111/j.1553-2712.2008.00339.x. Epub 2009 Jan 20. PMID 19154565
- [Background] Ryan DJ, O'Regan NA, Caoimh RO, Clare J, O'Connor M, Leonard M, McFarland J, Tighe S, O'Sullivan K, Trzepacz PT, Meagher D, Timmons S. Delirium in an adult acute hospital population: predictors, prevalence and detection. BMJ Open. 2013 Jan 7;3(1):e001772. doi: 10.1136/bmjopen-2012-001772. PMID 23299110